CLINICAL TRIAL: NCT07110168
Title: Robot-assisted Adrenalectomy, a Retrospective Single-center Study of 700 Procedures.
Brief Title: Robot-assisted Adrenalectomy, Feasibility and Results
Acronym: ROBADRE
Status: Active, not recruiting | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, NOMINE-CRIQUI Claire, Medical Doctor - Head of the endocrine surgery unit of the department of metabolic, endocrine and oncologic surgery, Central Hospital, Nancy, France
Other Study IDs: 2025PI122
Record Dates: First submitted 2025-07-31; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Adrenalectomy
Keywords: adrenalectomy; robotic surgery; robot-assisted surgery; transperitoneal adrenalectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients who underwent robot assisted adrenalectomy in University Hospital of Nancy: All patients who underwent a robotic adrenalectomy (all adrenal disease included) in the Department of Visceral,Metabolic and Oncologic surgery in University Hospital of Nancy between 01.01.2013 and 12.31.2025.

SUMMARY:
To date, laparoscopy is considered to be the gold standard technique for adrenalectomy. Robotic surgery is beginning to be used, but no series of more than 300 procedures has yet allowed the morbidity, benefits and learning curve of this technique to be assessed. Furthermore, the debate on the benefits of using robotic tools when performing adrenalectomies remains open. At Nancy University Hospital, we have been performing robotic procedures on 90% of our patients since 2009, and have seen a significant increase in patient numbers (currently between 80 and 90 per year).

In 2019, we published a series of 300 patients, describing the results of the technique.

Based on our clinical experience and the growing interest of the surgical community, we believe that describing our cohort of patients who have undergone robot-assisted surgery (estimated at 600 patients) is of unquestionable scientific interest.

In 2018, the American team at UCLA published a series of 640 laparoscopic adrenalectomies and examined the risk factors for complications following this surgery. Given the team's reputation and their publication in the leading surgical journal (JAMA Surgery), we used the same criteria for our data collection to make our results comparable.

This study aims to evaluate the risk factors for surgical complications after robotic adrenalectomy in a large retrospective series. Our aim is to demonstrate the safety and reliability of this technique and to identify patients at greatest risk of complications. This may encourage the adoption of the technique in other centres.

DETAILED DESCRIPTION:
Main objective:Evaluation of postoperative morbidity (Clavien-Dindo >2) 30 days after robot-assisted unilateral adrenalectomy

Secondary objective(s):

* Identify risk factors associated with the occurrence of complications after surgery. (patients characteristics, adrenal disease type)
* Determine the learning curve of robotic adrenalectomy considering surgical morbidity (Clavien Dindo>2)
* Determine the learning curve of robotic adrenalectomy considering operative time

Data collection:

PREOPERATIVE

Adrenal disease :

* Conn's adenoma
* Pheochromocytoma
* Cushing's adenoma
* Non-secreting adenoma
* Metastases (specify primary site: kidney, lung, skin)
* Virilising tumour
* Adrenal cancer (adrenocortical carcinoma)
* Haematological disorders
* Other

Patient characteristics:

* Age
* BMI
* ASA score
* Sex
* Comorbidity (Charleston score?)
* History of abdominal surgery/specify the procedure, noting whether it was laparoscopic or laparotomy
* History of adrenal surgery
* Genetic disease: NEM, VHL, etc.

Intra-operative data :

* Preoperative blood pressure
* Tumour laterality
* Surgeon
* Operative time
* Perioperative complications: bleeding, digestive tract injury, etc. ( using the KAARAFANI classification)
* Conversion to laparotomy and cause: adhesions, bleeding, digestive tract injury

Post-operative data :

* Length of hospital stay in days
* Morbidity: complications within 30 days after surgery according to Clavien-Dindo
* Mortality

ELIGIBILITY:
Inclusion Criteria:

* all patient who underwent unilateral robot-assisted adrenalectomy

Exclusion Criteria:

* bilateral adrenalectomy
* adrenalectomy by laparotomy
* partial adrenalectomy

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients who underwent robot-assisted adrenalectomy in Department of Visceral Metabolic and Oncologic surgery Department
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2025-05-30 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Morbidity after robotic adrenalectomy | from enrollment to 30 days after surgery
  evaluation of morbidity after robotic adrenalectomy in the 30 days after surgery using Clavien Dindo classification

SECONDARY OUTCOMES:
factors associated with clavien Dindo morbidity>2 | from enrollment to 30 days after surgery
  Using the data base, identification of factors related to patient or to adrenal disease associated with a higher post-operative morbidity
Learning curve | from enrollment to 30 days after surgery
  To determinate the learning curve of robotic adrenalectomy with a significant decrease of post-operative morbidity (number of cases)
Learning curve - operative time | from enrollment to 30 days after surgery
  To determinate the number of procedure necessary to significantly decrease the operative time

CONTACTS AND LOCATIONS:
Locations (1):
- Nomine-Criqui Claire, Nancy, Lorraine, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bihain F, Klein M, Nomine-Criqui C, Brunaud L. Robotic adrenalectomy in patients with pheochromocytoma: a systematic review. Gland Surg. 2020 Jun;9(3):844-848. doi: 10.21037/gs-2019-ra-05. PMID 32775278
- [Background] Giordano A, Balla A, Prosperi P, Morales-Conde S, Bergamini C. Robotic vs. Laparoscopic Adrenalectomy for Pheochromocytoma-A Systematic Review and Meta-Analysis. J Clin Med. 2025 May 29;14(11):3806. doi: 10.3390/jcm14113806. PMID 40507569
- [Background] Li X, Xiao S, Yu Y, Liu W, Xi H, Wang G, Zhou X. Robotic-assisted laparoscopic adrenalectomy (RARLA): What advantages and disadvantages compared to retroperitoneal laparoscopic adrenalectomy (RLA)? Front Endocrinol (Lausanne). 2023 Mar 2;14:1145820. doi: 10.3389/fendo.2023.1145820. eCollection 2023. PMID 36936166
- [Background] Chen Y, Scholten A, Chomsky-Higgins K, Nwaogu I, Gosnell JE, Seib C, Shen WT, Suh I, Duh QY. Risk Factors Associated With Perioperative Complications and Prolonged Length of Stay After Laparoscopic Adrenalectomy. JAMA Surg. 2018 Nov 1;153(11):1036-1041. doi: 10.1001/jamasurg.2018.2648. PMID 30090934
- [Background] Greilsamer T, Nomine-Criqui C, Thy M, Ullmann T, Zarnegar R, Bresler L, Brunaud L. Robotic-assisted unilateral adrenalectomy: risk factors for perioperative complications in 303 consecutive patients. Surg Endosc. 2019 Mar;33(3):802-810. doi: 10.1007/s00464-018-6346-2. Epub 2018 Jul 11. PMID 29998394